CLINICAL TRIAL: NCT00026663
Title: Collection of Blood, Fluid, Bone Marrow, Tumor, or Tissue Samples From Patients With Cancer or Normal Volunteers
Brief Title: Collection of Blood, Bone Marrow, Tumor, or Tissue Samples From Patients With Cancer to Study Drug Resistance
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000078; 00-C-0078; NCT00919529 (obsolete NCT alias)
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Renal Cell Carcinoma; Lung Carcinoma; Cervical Carcinoma
Keywords: Assays; Resistance; Biopsy Samples; Specimen Acquisition; Cancer Cells; Natural History
MeSH Terms: conditions — Carcinoma, Renal Cell; Lung Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Patients with cancer: Cancer patients providing tissue for research studies
- 2/Normal Volunteers: normal volunteers providing samples for research studies

SUMMARY:
This study will examine blood, bone marrow, tumor and tissue samples from patients with cancer to study tumor resistance to chemotherapy (drug treatment). Many patients with cancer improve initially with chemotherapy, but then have a disease relapse, after which their tumor no longer responds to treatment. Other patients tumors are drug-resistant from the start. The study will look for "resistance factors"-substances in blood and tissues that render tumors resistant to chemotherapy. The findings may provide information needed to develop methods of combating drug resistance.

Patients with cancer who are 18 years or older may be eligible for this study. Participants will have 40 milliliters (3 tablespoons) of blood drawn at the beginning of the study; additional samples will be obtained periodically during the course of treatment. A small sample of tumor or normal tissue will be taken from patients who undergo surgery or tumor biopsy (removal of a small piece of tumor) for medical reasons or as part of a research treatment protocol. Patients who do not require surgery or biopsy may be asked permission to obtain a tumor sample. Depending on the location of the tumor, this may be done by: 1) withdrawing bone marrow through a small needle; 2) removing fluid from the chest or abdomen; 3) removing a small tumor sample through a needle; or 4) removing the sample with a small incision into or around the tumor. These procedures will be done only if they are of low risk to the patient.

DETAILED DESCRIPTION:
Background:

Ongoing research in the Molecular Pharmacology Section, NCI, requires the availability of blood, fluid, bone marrow, tumor, hair follicle and tissue samples from patients with cancer. Resistance is the underlying cause of treatment failure, and may present as acquired or intrinsic drug resistance. Patients with cancer frequently present with chemotherapy-responsive disease, and undergo tumor response, only to eventually experience relapse, at which time the tumor may be refractory to further treatment. This is termed acquired drug resistance; while intrinsic resistance implies a cancer that is refractory from the outset. Diverse mechanisms of drug resistance have been described and are often dependent upon the particular drug under study.

Objectives:

To obtain blood, fluid, hair follicles, bone marrow, tumor and/or normal tissue samples that would allow development of assays for use in subsequent clinical trials.

Eligibility:

Patients with a prior diagnosis of malignancy, with advanced or refractory cancer will be evaluated in the GMB Clinic, NCI.

Participants may be on, or in the process of being evaluated for a research protocol. Participants may receive treatment on the standard care protocol.

Normal volunteers may enroll in the study.

Design:

Acquired samples will be recorded in the computerized data bank currently existing in the Molecular Pharmacology Section. No germline testing will be performed on any of the samples collected. Tests will be pilot studies relating to the Section s work on the biology of drug resistance and cell survival in cancer.

Sample collection for patients with cancer:

* Blood samples, fluid samples, or hair follicle samples may be collected at the initial visit, and at follow up visits.
* Tumor samples may be obtained by fine needle aspirate, by removal of pleural or peritoneal fluid, or by excisional biopsy, providing the tumor is accessible.
* Bone marrow aspirate, thoracentesis, and paracentesis may be performed.

Normal volunteers may enroll in the study for collection of blood, fluid, and/or hair follicle samples.

Examples of the types of studies to be performed with biopsies will be drug resistance gene expression assays, with the goal of demonstrating the utility of the assay in participant samples.

Evaluation of methods to detect drug resistance proteins and genes will be explored, including Northern blot, immunoblot, polymerase chain reaction assay, and RNA in situ hybridization. With whole blood, we may evaluate the presence of dye transport in an ex vivo assay, for example, using inhibitors of ABCG2. Evidence of drug accumulation or DNA damage may be sought in participant mononuclear cells or in hair follicle samples.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participants 18 years of age and older are eligible.
  2. Participants must have a performance status of ECOG 0, 1, 2, or 3 for admission to this protocol.
  3. Participants with malignancy are eligible.
  4. Participants requiring a surgical procedure for any medical indication can be included on study.
  5. Participants requiring biopsy or any procedure for any medical indication can be included on study.
  6. Participants not requiring biopsy for a medical indication can be included on the study solely for the purpose of obtaining research samples, including blood, pleural fluid, or peritoneal fluid, or biopsy samples. No radiology tests will be used in the procedure to collect a sample that would not be otherwise used for an appropriate medical indication.
  7. Normal volunteers 18 years of age and older are eligible to enroll. Normal volunteers must be willing to sign informed consent and must be willing to provide samples to be used for research.

EXCLUSION CRITERIA:

1. Pregnant individuals will not be eligible due to potential risks to the fetus associated with radiologic procedures required for biopsy.
2. Children will not be eligible because of potential risks from complications due to procedures involved in obtaining the biopsies.
3. Normal volunteers with a history of a clotting disorder may not enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with malignancy requiring a surgical procedure or biopsy for any medical indication. Healthy volunteers not requiring biopsy for a medical indication.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2000-08-09 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
To obtain specimens to develop assays | End of study
  Obtain sufficient number of samples for a given test.

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-C-0078.html